CLINICAL TRIAL: NCT03755557
Title: Demonstration of Therapeutic Equivalence/Non-inferiority as Well as Early Onset of Action of the Novel Water-soluble Budesonide Nasal Spray (Budesolv 10) Compared With Marketed Rhinocort® Aqua 64 in Patients Suffering From Grass Pollen Induced Allergic Rhinitis
Brief Title: Demonstration of Equivalence and Early Onset of a Novel Anti-allergic Nasal Spray Compared to Marketed Nasal Spray
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Marinomed Biotech AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BDS_18_01; 2018-001324-19 (EudraCT Number)
Record Dates: First submitted 2018-11-21; First posted 2018-11-28 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Allergic Rhinitis; Allergic Conjunctivitis; Hayfever
Keywords: budesonide; allergic rhinitis; allergic rhinoconjuntivitis; allergen exposure chamber; onset of action; therapeutic equivalence; total nasal symptom score; hayfever; glucocorticosteroids; nasal congestion; Vienna Challenge Chamber; Carragelose; Carrageenan; Iota-Carrageenan
MeSH Terms: conditions — Rhinitis, Allergic; Conjunctivitis, Allergic; Rhinitis, Allergic, Seasonal; Nasal Obstruction | interventions — Budesonide

STUDY DESIGN:
Intervention Model Description: 3-way crossover, randomized, prospective, placebo-controlled, double blinded study in a validated allergen exposure chamber setting using grass pollen allergen
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The visual aspects of the three treatment arms are identical. Identification of the treatment is achieved via a randomization code.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Application of a placebo nasal spray once daily for 8 days Nasal Sprays
  Interventions: Other: Placebo
- Rhinocort (Active Comparator): Nasal Sprays Application of "Rhinocort Aqua 64 micrograms, nasal spray" once daily for 8 days. Daily dosage 256 µg/d
  Interventions: Drug: Rhinocort
- Budesolv (Experimental): Application of a Budesolv 10 micrograms, nasal spray once daily for 8 days. Daily dosage 40 µg/d Nasal Sprays
  Interventions: Drug: Budesolv

INTERVENTIONS:
Drug: Rhinocort — Application of a nasal spray
  Other Names: Budesonide
  Arms: Rhinocort
Drug: Budesolv — Application of a nasal spray
  Other Names: Budesonide
  Arms: Budesolv
Other: Placebo — Application of a nasal spray
  Other Names: buffered saline
  Arms: Placebo

SUMMARY:
Intranasal corticosteroids are accepted as safe and effective first-line therapy for allergic rhinitis, especially in treatment of persistent symptoms.

Budesonide, a non-halogenic glucocorticoid, is widely used in the management of inflammatory mucosal diseases like chronic obstructive pulmonary disease, asthma and allergic rhinitis. It is a highly fat-soluble substance with low water solubility and is presented as dispersion in marketed nasal sprays, like Rhinocort aqua 64. The maximum therapeutic efficacy of Rhinocort aqua is obtained after an application period of 7 to 14 days. In Budesolv, the solubility of budesonide is considerably increased suggesting that the same therapeutic efficacy can be reached with a lower dose. Better bioavailability of the dissolved drug promise an earlier onset of therapeutic efficacy. The current trial is undertaken to demonstrate these two effects. Subjects suffering from grass pollen allergic rhinitis will be challenged with grass pollen in a challenge chamber.

Allergic subjects will be treated with two actuations (50 μl) of respective study treatment into each nostril once daily for 8 days. The total daily budesonide dose will be 40 μg per subject for Budesolv 10 and 256 μg per subject for Rhinocort® aqua 64. The primary objective of the study is to show non-inferiority of Budesolv 10 to Rhinocort® aqua 64. On day 8 grass pollen allergic patients will be challenged with grass pollen over a period of 6 hours and subjective nasal symptoms (congestion, sneezing, itching, rhinorrhea) as well as objective symptoms (nasal airflow, nasal secretion) will be assessed every 15 minutes.

The second objective of the trial is to demonstrate an early on-set of therapeutic efficacy of Budesolv 10 compared to Rhinocort aqua. On day 1, grass pollen allergic patients will be challenged with grass pollen allergen in the challenge chamber over a period of 6 hours. After 1 hour 45 minutes, patients will receive their first dosage of the respective nasal spray treatment. During the 6 hour grass pollen challenge, subjective and objective endpoints will be measured every 15 minutes.

To eliminate an individual bias based on expectations, the effect and onset of action is also compared to the effects of a suitable placebo. The same set of study participants will receive all three interventions in three consecutive treatment periods.

DETAILED DESCRIPTION:
This is a randomized, placebo controlled, three way cross over, double-blind, single site trial in adult subjects (18 years of age and older) who demonstrate grass specific Immunglobulin E (IgE) reactivity and have a history of grass pollen induced allergic rhinitis/rhinoconjunctivitis with or without controlled asthma. In the cross-over setting three treatments, namely placebo, Budesolv 10 or Rhinocort® aqua 64 will be evaluated.

The primary objective of the trial is to demonstrate therapeutic equivalence/non-inferiority between Budesolv 10 and Rhinocort® aqua 64, a marketed comparator containing the same compound (budesonide), in patients suffering from grass pollen induced allergic rhinitis/rhinoconjunctivitis with or without controlled asthma on day 8 of treatment. A placebo group will be introduced to show effectiveness of treatment and hence validate the trial design.

The evaluation will be based on the assessment of rhinitis symptoms during grass pollen challenge performed in the Vienna Challenge Chamber (environmental exposure chamber).

Secondary objective of the trial is the early onset of action of Budesolv 10 compared to Rhinocort® aqua 64, determined on day one of treatment.

Visit 1 + 2 - Screening + Inclusion period:

Subjects will be screened for appropriate allergic response. A total nasal symptom score (TNSS) of at least 6 points out of 12 within the first two hours in the grass pollen challenge chamber is required to be included into the study.

Visit 3 + 5 + 7 / "day 1":

Eligible subjects will be randomly assigned to one of the three treatment arms (fully blinded) in the order of their screening numbers assigned at visit 1. Subjects will enter the study site about one hour ahead of the start of allergen provocation. After positive completion of all study relevant assessments, subjects enter the grass pollen challenge chamber for subjective and objective assessments for a period of 6 hours. One hour forty-five minutes after entry, the first treatment will be applied.

The subjective nasal symptom score will be recorded every fifteen minutes during a 6-hour allergen exposure challenge. Every hour rhinomanometry will be performed to objectively evaluate the respiratory function of the nose. Additional rhinomanometry will be performed at two hours 30 minutes after entry. Subjects will continue treatment with two actuations into each nostril once a day until day 7.

Visit 4 + 6 + 8 / "day 8":

On day 8 of their respective treatment block, subjects will enter the study site about two hours before provocation will start. Subjects will take their last treatment dosage approximately one hour before entering the challenge chamber. The study medication device will be returned to study site staff for external analytical evaluations after usage (in-use-stability test). After receiving their last treatment dose and shortly before entering the challenge chamber, baseline symptom score will be assessed. Like on day one, subjects will be provoked for 6 hours with grass pollen allergens. Subjective symptom scores will be recorded every fifteen minutes, and rhinomanometry will be performed every hour during the challenge.

Between the respective study treatments, a wash-out period of at least 20 days must be adhered to allowing complete dissipation of the previous treatment. After the wash-out period, subjects change to the next treatment block in the sequence. During the entire trial, subjects will be asked to monitor for adverse events (AEs), and they will record the use of concomitant medications on the provided form. Female subjects of child-bearing potential will complete a urine pregnancy test in the course of all visits.

Following parameters will be assessed:

* Subjective symptom score (nasal, ocular, respiratory) during a grass pollen challenge lasting for 6 hours - every 15 minutes Active anterior rhinomanometry (AAR) - every 60 minutes, additional measurement on day 1 at 2:30 after entry.
* Lung function tests using regular spirometry for FEV1 and FVC - every 120 minutes
* Nasal secretion weight - every 30 minutes
* Physical examination - at Screening and Follow up
* Vital signs - every visit, pre- and post-challenge
* Safety laboratory assessments: Complete blood count with differential, blood chemistry, liver function, urine dipstick test - at screening and last treatment visit, serology at screening and drug abuse test on investigator's decision
* Skin Prick Test with skin prick test solution (Manufacturer Allergopharma) - at Screening or within the previous 6 months
* Specific CAP analysis (g6) - at Screening or within the previous 6 months
* ECG - at screening and Follow up
* Adverse events - throughout the study
* Concomitant medication - throughout the study One week after the final provocation session, subjects will complete the trial after their follow up visit. Validated methods of data collection, analysis, and evaluation will be used for the trial.

The trial endpoints are listed below:

Primary efficacy endpoint:

The primary efficacy endpoint will be the mean 'Total Nasal Symptom Score' (TNSS), calculated as the baseline adjusted mean of TNSS measured at 17 time points (every 15 minutes) during the grass pollen allergen exposure challenge from time point 2 to 6 hours on day 8.

The TNSS is the sum of the symptoms "nasal congestion", "rhinorrhea", "itchy nose" and "sneezing". Each individual symptom will be scored on a 4-point categorical scale from 0-3 (where "0"= none "1"=mild "2"=moderate "3"=severe).

Key Secondary efficacy endpoint:

Time point when onset of action can be observed.

Additional secondary efficacy endpoints:

* Nasal airflow: will be assessed every hour during the six hour grass pollen allergen exposure challenge
* Nasal secretion: will be assessed every 30 minutes during the six-hour grass pollen allergen exposure challenge. Additional rhinomanometry will be done on day 1 at 2:30 h after entry in the challenge chamber
* Total ocular symptom score (TOSS) is the sum of the symptoms "ocular itching", "redness", "watery eyes".
* Total asthma symptom score (TASS) is the sum of the symptoms "cough", "wheeze", "dyspnea".

Each individual symptom of TOSS and TASS will be scored on a 4-point categorical scale from 0-3 (where "0"= none "1"=mild "2"=moderate "3"=severe). TOSS and TASS will be assessed every 15 minutes during the six-hour grass pollen allergen exposure challenge.

Safety endpoints:

* Adverse events (AEs)
* Safety laboratory
* ECG
* Spirometry (FeV1, FVC)

ELIGIBILITY:
Inclusion criteria

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

* Written informed consent obtained before any trial related procedures are performed
* Healthy male or female subjects aged 18 years or older
* Female subjects of child-bearing potential must have a negative pregnancy test and be willing to practice appropriate contraceptive methods until the end of treatment visit
* A documented clinically relevant allergic history of moderate to severe SAR to grass pollen for the previous two years
* Subjects exhibit a moderate to severe response to approximately 1500 grass pollen grains/m3 within the first 2 hours in the Vienna Challenge Chamber, which is defined as total nasal symptom score (TNSS) of at least 6 (out of 12) using standard VCC grass pollen allergen mixture. Nasal symptom score is the sum of "nasal congestion", "rhinorrhea", "itchy nose" and "sneezing", each of which have been scored on a categorical scale from 0 to 3.
* Positive Skin Prick Test (SPT) response (wheal diameter at least 3 mm larger than diluent control) to grass pollen SPT solutions (standard Allergopharma) at screening or within the last 6 months prior to study start.
* Positive serum specific IgE against recombinant major allergen components of the used grass pollen (specific CAP IgE ≥0.70 kU/L) at screening or within the last 6 months prior to study start.
* Patients with a body weight of ≥ 50kg and a body mass index within the range of 19-30kg/m2.
* Non-smoking subjects (smoked <10 packs years in their lifetime and had not smoked in the last 6 months)
* Asthma patients only if the asthma condition is mild or intermittent, and if those are not treated with steroids
* Subject has a forced expiratory volume in 1 second (FEV1) of at least 80% of predicted value (ECCS) at the screening.
* Subject is capable of understanding the study procedures and potential risks associated with the study, and voluntarily agrees to participate by giving written informed consent.
* Subject is able to adhere to dose and visit schedules.
* Subject is able to read, understand and complete questionnaires and diaries.

Exclusion Criteria

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Pregnant, lactating or sexually active women with childbearing potential who are not using a medically accepted birth control method (pregnancy to be controlled by a pregnancy dipstick test).
* A clinical history of uncontrolled asthma within 3 months prior to screening.
* Subjects with asthma requiring treatment with inhaled corticosteroids on a regular basis judged by the investigator.
* Previous successful immunotherapy to grass pollen, a grass pollen allergen or a cross-reacting allergen within the past 3 years.
* Ongoing treatment with any allergen-specific immunotherapy product.
* Subjects with a current oral candidiasis infection or treatment for oral candidiasis during the last 30 days before starting the study.
* Subjects with history of tuberculosis.
* Subjects with any fungal/viral/bacterial respiratory or systemic infections during the last 30 days.
* Symptoms of or treatment for upper respiratory tract infection, acute sinusitis, acute otitis media or other relevant infectious process at randomization.
* Clinically relevant nasal polyps, medical history of paranasal sinus surgery and/or medical history of surgery of nasal turbinates judged by the investigator.
* Subjects with glaucoma or a family history of glaucoma.
* Subjects using any ophthalmic steroids during the last 30 days.
* Subjects treated with nasal, inhaled or systemic steroids during the last 30 days.
* History of anaphylaxis with cardiorespiratory symptoms (immunotherapy, exercise induced, food allergy, drugs or an idiopathic reaction).
* Any clinically relevant chronic disease judged by the investigator.
* Systemic disease affecting the immune system judged by the investigator.
* Use of an investigational drug within 30 days/5 half-lives of the drug (which ever longest) prior to screening.
* History of allergy, hypersensitivity or intolerance to any ingredients of the IMP.
* History of alcohol or drug abuse.
* Being immediate family of the investigator or trial staff, defined as the investigator's/staff's spouse, parent, child, grandparent or grandchild.
* Subjects with previous SAR that has proven unresponsive to steroid therapy.
* Subjects treated with leukotriene antagonists (1 month before study start), long-lasting anti-histamines, like cetirizine, fexofenandine, loratadine, desloratadine, hydroxyzine (5 to 10 days before study start), mast cell stablizier (2 weeks before study start) or nasal decongestant (3 days before study start).
* Subjects with an acute or chronic sinusitis judged by the investigator.
* Subjects with hypersensitivity to corticosteroids judged by the investigator.
* Subjects with ocular herpes simplex infections.
* Subjects with cataracts and with cataract history.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-05 (Actual)

PRIMARY OUTCOMES:
Total Nasal Symptom Score | 2 - 6 hours of allergen challenge
  subjective compound score evaluating "nasal congestion", "rhinorrhea", "itchy nose" and "sneezing" from "0" (absent) to "3" (severe). The sum of sub-scores is reported as total nasal symptom score (0 - 12)

SECONDARY OUTCOMES:
Total Ocular Symptom Score | 2 - 6 hours of allergen challenge
  subjective compound score evaluating "ocular itching", "redness", "watery eyes" from "0" (absent) to "3" (severe). The sum of sub-scores is reported as total ocular symptom score (0 - 9)
Total Asthma Symptom Score | 2 - 6 hours of allergen challenge
  subjective compound score evaluating "cough", "wheeze", "dyspnea" from "0" (absent) to "3" (severe). The sum of sub-scores is reported as total asthma symptom score (0 - 9)
Nasal airflow | 0 - 6 hours of allergen challenge
  Rhinomanometry
Nasal secretion | 0 - 6 hours of allergen challenge
  tissue weight

CONTACTS AND LOCATIONS:
Overall Officials: Eva E Prieschl-Grassauer, PhD, Study Chair — Marinomed Biotech AG
Locations (1):
- Vienna Challenge Chamber, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murdoch RD, Bareille P, Ignar D, Miller SR, Gupta A, Boardley R, Zieglmayer P, Zieglmayer R, Lemel P, Horak F. The improved efficacy of a fixed-dose combination of fluticasone furoate and levocabastine relative to the individual components in the treatment of allergic rhinitis. Clin Exp Allergy. 2015 Aug;45(8):1346-55. doi: 10.1111/cea.12556. PMID 25900517